CLINICAL TRIAL: NCT07172152
Title: Improving Minority Health Through Biofeedback and Stress Reduction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Amelia Saul, PhD, CTRS, BCB (Other)
Collaborators: University of Puerto Rico (Other)
Responsible Party: Sponsor-Investigator, Amelia Saul, PhD, CTRS, BCB, Assistant Teaching Professor, Florida International University
Organization: Florida International University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RB-23-0122-AM02
Record Dates: First submitted 2025-09-08; First posted 2025-09-15 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-09

CONDITIONS: Cardiovascular Disease Risk Reduction; Chronic Stress; Anxiety; Emotional Regulation; Hypertension Prevention; Health Disparities
Keywords: Heart Rate Variability; Biofeedback; Stress Reduction; Anxiety Management; Cardiovascular Health; Emotional Regulation; Preventative Health; Mind-Body Intervention
MeSH Terms: conditions — Anxiety Disorders; Emotional Regulation

STUDY DESIGN:
Intervention Model Description: This study follows a randomized controlled trial (RCT) design with a parallel assignment of participants into two groups:
  Intervention Group: Receives a four-week HRV biofeedback training. Control Group: No intervention, continues with usual activities.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HRV Biofeedback Intervention Group (Experimental): Participants in this group will receive HRV biofeedback training for four weeks. They will attend five sessions: an initial baseline session, three weekly check-in sessions, and a final post-intervention assessment.
  HRV biofeedback training will utilize an app that will provide guidance to participants to follow a pacer and breathe for 10 minutes and feedback will be provided.
  Interventions: Behavioral: HRV Biofeedback Training
- Control Group (No Intervention): Participants in this group will complete baseline and post-study assessments but will not receive the HRV biofeedback intervention. They will continue their usual daily activities without specific stress management training.

INTERVENTIONS:
Behavioral: HRV Biofeedback Training — Participants will be trained to use HRV biofeedback through paced breathing exercises (6 breaths per minute) twice daily over a four-week period.
  Other Names: HRVB
  Arms: HRV Biofeedback Intervention Group

SUMMARY:
This study aims to evaluate the effectiveness of a four-week heart rate variability (HRV) biofeedback intervention to improve physiological stress response, emotion regulation, and anxiety-related symptoms in young ethnic minority adults with a family history of cardiovascular disease (CVD). Participants will be randomly assigned to either an intervention group, where they will engage in guided paced breathing exercises, or a control group, which will follow standard conditions without the intervention.

The study consists of five sessions, including an initial assessment, three weekly check-in sessions, and a final post-intervention assessment. Participants will practice paced breathing at home and attend brief in-lab sessions to track progress. Physiological and psychological measures, such as HRV, GSR, BP, anxiety levels, and responses to the Socially Evaluated Cold Pressor Test (SECPT), will be used to assess outcomes. Findings from this study may provide insights into accessible, non-invasive stress management interventions to mitigate CVD risk in high-risk populations.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is the leading cause of death in the United States, disproportionately affecting racial and ethnic minority populations. Chronic stress has been identified as a significant risk factor for CVD, yet few interventions address stress reduction as a preventative measure. This study investigates whether HRV biofeedback training can serve as an effective, non-pharmacological intervention to improve stress resilience and reduce risk factors associated with CVD.

ELIGIBILITY:
Inclusion Criteria:

* Adults
* Age 18 to 35 years
* Cognitively intact to follow instructions
* English-speaking
* Family history of cardiovascular disease.

Exclusion Criteria:

* Cognitive impairments that inhibit understanding instruction
* Current diagnosis of hypertension that is controlled with prescribed medication
* Previously receiving biofeedback training
* Having a severe medical condition (e.g., pacemaker, cardiac arrhythmia, hypertension, diabetes)
* Being actively psychotic
* Having a neurological condition (e.g., Parkinson's disease) that would complicate the interpretation of physiological data
* Patients currently taking medications such as MAOIs, alpha/beta-blockers, or withdrawal or maintenance medications (e.g., Librium, methadone) are excluded due to their potential to affect the HRV data

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Heart Rate Variability Improvement | 4 weeks
  HRV will be assessed using the OptimalHRV sensor to determine improvements in autonomic regulation and stress resilience.
State Anxiety Reduction (Beck Anxiety Inventory - BAI) | 4 weeks
  Changes in self-reported state anxiety levels will be assessed before and after the HRV biofeedback intervention using the Beck Anxiety Inventory (BAI). The BAI is a 21-item self-report questionnaire designed to measure anxiety severity. Each item is scored on a 4-point Likert scale ranging from 0 ("Not at all") to 3 ("Severely-it bothered me a lot"), resulting in a total score ranging from 0 to 63. Higher scores indicate greater levels of anxiety, while lower scores indicate reduced anxiety.
Stress Resilience Under Acute Stress (Socially Evaluated Cold Pressor Test - SECPT) | 4 weeks
  The Socially Evaluated Cold Pressor Test (SECPT) will be used to measure changes in both self-reported and physiological stress responses to an acute stressor. Self-reported distress will be measured using a Visual Analog Scale, a 0-10 scale where 0 = no pain and 10 = worst possible pain. Higher scores indicate worse outcomes (greater distress). Emotional response will be measured using the Self-Assessment Manikin (SAM), which assesses valence, arousal, and dominance on a 5-point pictorial scale. Scores are coded such that higher valence = more positive affect, higher arousal = greater activation, and higher dominance = greater sense of control.

SECONDARY OUTCOMES:
Blood Pressure | 4 weeks
  Change in systolic and diastolic blood pressure.
Galvanic Skin Response (GSR; Electrodermal Activity) | 4 weeks
  Change in skin conductance level (SCL) and response frequency during stress and recovery tasks.

CONTACTS AND LOCATIONS:
Overall Officials: Amelia D Saul, PhD, Principal Investigator — Florida International University
Locations (1):
- Florida International University, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Shaffer F, Ginsberg JP. An Overview of Heart Rate Variability Metrics and Norms. Front Public Health. 2017 Sep 28;5:258. doi: 10.3389/fpubh.2017.00258. eCollection 2017. PMID 29034226
- [Result] Bolin LP, Saul AD, Bethune Scroggs LL, Horne C. A pilot study investigating the relationship between heart rate variability and blood pressure in young adults at risk for cardiovascular disease. Clin Hypertens. 2022 Jan 15;28(1):2. doi: 10.1186/s40885-021-00185-z. PMID 35031077